CLINICAL TRIAL: NCT05441059
Title: Evaluation of Real World Use of Nucala in Severe Asthma Patients From the Severe Heterogenous Asthma Research Patient-centred Collaboration (SHARP)
Brief Title: Use of Nucala in Severe Asthma
Acronym: UNISA
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 212821
Record Dates: First submitted 2022-06-21; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Asthma Severe Persistent Uncontrolled
MeSH Terms: interventions — mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with mepolizumab: Patients treated with mepolizumab
  Interventions: Drug: Mepolizumab 100 MG

INTERVENTIONS:
Drug: Mepolizumab 100 MG — Treatment with mepolizumab for severe asthma

SUMMARY:
The Severe Heterogeneous Asthma Research collaboration, Patient-centred (SHARP) is set up to harmonise severe asthma management across Europe and unravel underlying heterogeneity in a patient-centred way. Using data from national registries included in the SHARP network, this study aims to evaluate real-world use of Nucala, describe characteristics of patients prescribed with Nucala and evaluate the effectiveness of Nucala in clinically relevant endpoints.

DETAILED DESCRIPTION:
The global prevalence of asthma is approximately 358 million people, of which an estimated 30 million patients live in Europe. Severe asthma is defined as asthma requiring treatment according to GINA steps 4-5 and is estimated to occur in 5-10% of the total asthma population (Chung 2014). Asthma and severe asthma are heterogeneous, and while there are a range of classifications, one such schema classified asthma as: (1) eosinophilic, (2) neutrophilic, (3) mixed, or (4) paucigranulocytic.

NUCALA (mepolizumab) is an IL-5 antagonist monoclonal antibody that was approved by the European commission in 2015 for add-on maintenance treatment of adult patients with severe refractory eosinophilic asthma. The license was expanded to paediatric patients (6-17 years old) in August 2018. Clinical efficacy was evaluated in multiple randomized, double-blind clinical trials. In the DREAM trial (NCT01000506), the rate of clinically significant exacerbations was 2.40 per patient per year among patients receiving placebo versus 1.24 in the 75 mg IV mepolizumab group, a 48% (95% CI 31-61%) reduction. In the MENSA trial (NCT01691521), the rate of clinically significant exacerbations was 1.74 per patient per year among patients receiving placebo versus 0.83 in the sub-cutaneous 100 mg mepolizumab group, a 53% (95% CI 36-65%) reduction. Furthermore, in the SIRIUS trial (NCT01691508), the median daily prednisone dose at weeks 20-24 was 10.0 mg among patients receiving placebo versus 3.1 mg for patients receiving 100 mg of mepolizumab and mepolizumab provided a 2.39 (95% CI 1.25-4.56) times greater odds for a reduction in oral glucocorticoid dose from baseline in the mepolizumab group compared with placebo. Additionally, the MUSCA trial (NCT02281318) found that mepolizumab significantly improved health-related quality of life in patients with severe eosinophilic asthma.

The high internal validity of the randomized clinical trials has allowed the treatment efficacy of Nucala to be reliably determined in patients with severe eosinophilic asthma. However, the strict inclusion and exclusion criteria which are necessary in clinical trials produce data from a selected, homogeneous population which may not be representative of the wider population who may receive treatments in routine practice.

Real world evaluation of mepolizumab use will help in understanding characteristics of patients from different European countries receiving these therapies, treatment patterns, and effectiveness on clinical endpoints as limited information exists in real world settings in Europe following the availability of mepolizumab to patients.

The Severe Heterogeneous Asthma Research collaboration, Patient-centred (SHARP) is set up to harmonise severe asthma management across Europe and unravel underlying heterogeneity in a patient-centred way. Using data from national registries included in the SHARP network, this study aims to evaluate real-world use of Nucala, describe characteristics of patients prescribed with Nucala and evaluate the effectiveness of Nucala in clinically relevant endpoints.

ELIGIBILITY:
Inclusion Criteria:

1) Initiated on mepolizumab for treatment of asthma.

Exclusion Criteria:

1) Participation in an interventional clinical trial in which the treatment regimen and/or monitoring is dictated by a protocol in the study observation period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be selected from all patients who meet the criteria for inclusion in individual registries severe asthma registries. Within this severe asthma population, the study sample will include all patients who received at least one dose of mepolizumab.
Sampling Method: Probability Sample
Enrollment: 2100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The change from baseline rate of annualized asthma exacerbations 1 year after initiation with mepolizumab | 1 year
  The change from baseline rate of annualized asthma exacerbations 1 year after initiation with mepolizumab
The change from baseline maintenance oral corticosteroid dose (mg/day, predinisone equivalents) 1 year after initiation with mepolizumab | 1 year
  The change from baseline maintenance oral corticosteroid dose (mg/day, predinisone equivalents) 1 year after initiation with mepolizumab

SECONDARY OUTCOMES:
Clinical and patient reported measures of asthma control (ACT and/or ACQ) in the periods before and after initiation with mepolizumab | 1 year
  Clinical and patient reported measures of asthma control (ACT and/or ACQ) in the periods before and after initiation with mepolizumab
The change from baseline measures of healthcare utilisation (number of hospitalisations and emergency department visits) 1 year after initiation with mepolizumab | 1 year
  The change from baseline measures of healthcare utilisation (number of hospitalisations and emergency department visits) 1 year after initiation with mepolizumab
Proportion of patients who stop mepolizumab after 1 year after initiation | 1 year
  Proportion of patients who stop mepolizumab after 1 year after initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: No
IPD is not available in this study due to the federated analysis of data.

REFERENCES:
- [Background] Simpson JL, Scott R, Boyle MJ, Gibson PG. Inflammatory subtypes in asthma: assessment and identification using induced sputum. Respirology. 2006 Jan;11(1):54-61. doi: 10.1111/j.1440-1843.2006.00784.x. PMID 16423202
- [Background] Pavord ID, Korn S, Howarth P, Bleecker ER, Buhl R, Keene ON, Ortega H, Chanez P. Mepolizumab for severe eosinophilic asthma (DREAM): a multicentre, double-blind, placebo-controlled trial. Lancet. 2012 Aug 18;380(9842):651-9. doi: 10.1016/S0140-6736(12)60988-X. PMID 22901886
- [Background] Taille C, Chanez P, Devouassoux G, Didier A, Pison C, Garcia G, Charriot J, Bouee S, Gruber A, Pribil C, Bourdin A, Humbert M. Mepolizumab in a population with severe eosinophilic asthma and corticosteroid dependence: results from a French early access programme. Eur Respir J. 2020 Jun 25;55(6):1902345. doi: 10.1183/13993003.02345-2019. Print 2020 Jun. PMID 32241829
- [Background] Ortega HG, Liu MC, Pavord ID, Brusselle GG, FitzGerald JM, Chetta A, Humbert M, Katz LE, Keene ON, Yancey SW, Chanez P; MENSA Investigators. Mepolizumab treatment in patients with severe eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1198-207. doi: 10.1056/NEJMoa1403290. Epub 2014 Sep 8. PMID 25199059
- [Background] Harrison T, Canonica GW, Chupp G, Lee J, Schleich F, Welte T, Valero A, Gemzoe K, Maxwell A, Joksaite S, Yang S, Howarth P, Van Dyke MK. Real-world mepolizumab in the prospective severe asthma REALITI-A study: initial analysis. Eur Respir J. 2020 Oct 15;56(4):2000151. doi: 10.1183/13993003.00151-2020. Print 2020 Oct. PMID 32817259
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Chupp GL, Bradford ES, Albers FC, Bratton DJ, Wang-Jairaj J, Nelsen LM, Trevor JL, Magnan A, Ten Brinke A. Efficacy of mepolizumab add-on therapy on health-related quality of life and markers of asthma control in severe eosinophilic asthma (MUSCA): a randomised, double-blind, placebo-controlled, parallel-group, multicentre, phase 3b trial. Lancet Respir Med. 2017 May;5(5):390-400. doi: 10.1016/S2213-2600(17)30125-X. Epub 2017 Apr 5. PMID 28395936
- [Background] Bel EH, Wenzel SE, Thompson PJ, Prazma CM, Keene ON, Yancey SW, Ortega HG, Pavord ID; SIRIUS Investigators. Oral glucocorticoid-sparing effect of mepolizumab in eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1189-97. doi: 10.1056/NEJMoa1403291. Epub 2014 Sep 8. PMID 25199060